CLINICAL TRIAL: NCT05856136
Title: Investigation of the Effects of Opioid Exposure on the Ability of the Diaphragm Muscle to Generate Higher Force Behaviors
Brief Title: A Study to Investigate of the Effects of Opioid Exposure on the Ability of the Diaphragm Muscle
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Carlos B Mantilla, MD, PhD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20-007084; R21DA055848 (NIH)
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Respiratory Function Loss; Respiratory Complication
Keywords: elastography; ultrasound
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ultrasound Shear Wave Elastography Examination - Lower (Experimental): Subjects identified as being administered low dose opioids during an elective lower extremity orthopedic surgery per standard of care will undergo an ultrasound shear wave elastography examination while performing different breathing techniques.
  Interventions: Drug: Fentanyl Injection
- Ultrasound Shear Wave Elastography Examination - Mid (Experimental): Subjects identified as being administered mid dose opioids during an elective lower extremity orthopedic surgery per standard of care will undergo an ultrasound shear wave elastography examination while performing different breathing techniques.
  Interventions: Drug: Fentanyl Injection
- Ultrasound Shear Wave Elastography Examination - Higher (Experimental): Subjects identified as being administered higher dose opioids during an elective lower extremity orthopedic surgery per standard of care will undergo an ultrasound shear wave elastography examination while performing different breathing techniques.
  Interventions: Drug: Fentanyl Injection

INTERVENTIONS:
Drug: Fentanyl Injection — Three different fentanyl doses (used for sedation) will be evaluated on their effects on shear wave elastography (SWE) and breathing

SUMMARY:
The purpose of this study is to evaluate opioid dose effects on the ability of the diaphragm muscle to generate higher force behaviors.

ELIGIBILITY:
Inclusion Criteria:

- Adult male and female patients undergoing lower extremity orthopedic surgery at the study institutions (St. Mary Hospital and Rochester Methodist Hospital within the Mayo Clinic Rochester hospital system).

Exclusion Criteria:

* Patients who refuse research participation.
* Patients who are pregnant.
* Patients with known pulmonary pathology (COPD, asthma requiring routine treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in shear wave speed | Baseline, 1 hour
  Measured by the ultrasound elastography of the diaphragm muscle reported in m/sec

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Mantilla, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No